CLINICAL TRIAL: NCT05136638
Title: A Randomized Controlled Comparative Trial of Digital Cognitive Behavioral Therapy for Insomnia (dCBTi): Comparing Efficacy and Adherence to dCBTi With Virtual and Human Coaching
Brief Title: dCBTi With and Without Coaching Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Wai Sze, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA210458
Record Dates: First submitted 2021-11-03; First posted 2021-11-29 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Insomnia
Keywords: Digital intervention; Cognitive Behavioral Therapy for Insomnia; Treatment efficacy; Treatment adherence
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All outcome measures will be administered via online surveys
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Digital Sleep Hygiene and Self-Monitoring Control (Active Comparator): Participants assigned to this condition will receive an app to track sleep and offers sleep hygiene recommendations
  Interventions: Behavioral: Sleep Hygiene and Self-Monitoring Control
- dCBTi without coaching (Experimental): Participants assigned to this condition will receive a 6-module digital cognitive behavioral therapy for insomnia (dCBTi) with no coaching support
  Interventions: Behavioral: dCBTi
- dCBTi with virtual coaching (Experimental): Participants assigned to this condition will receive a 6-module digital cognitive behavioral therapy for insomnia (dCBTi) with a virtual coach in the form of a text-based force-choice conversation coach. The virtual coach will check participants' understanding of the treatment materials and lead them to come up with action plans to implement CBTi strategies.
  Interventions: Behavioral: dCBTi; Behavioral: Virtual coaching
- dCBTi with non-therapist coaching support (Experimental): Participants assigned to this condition will receive a 6-module digital cognitive behavioral therapy for insomnia (dCBTi) with the virtual coach. They will get additional support from a non-therapist support person who provides support after modules 1, 3, and 6 to address any questions or concerns.
  Interventions: Behavioral: dCBTi; Behavioral: Virtual coaching; Behavioral: Non-therapist coaching
- dCBTi with therapist coaching support (Experimental): Participants assigned to this condition will receive a 6-module digital cognitive behavioral therapy for insomnia (dCBTi) with the virtual coach. They will get additional support from a clinical psychology trainee who provides therapeutic support that aims to enhance the usage of CBTi treatment strategies.
  Interventions: Behavioral: dCBTi; Behavioral: Virtual coaching; Behavioral: Therapist coaching

INTERVENTIONS:
Behavioral: dCBTi — The dCBTi adopts a multi-module approach, consisted of 6 weekly modules including psychoeducational on sleep, insomnia, sleep hygiene, sleep restriction and prescription, stimulus control, relaxation and worry time, cognitive restructuring, and relapse prevention. In each module, participants will watch short videos to learn strategies to improve their sleep.
  Arms: dCBTi with non-therapist coaching support; dCBTi with therapist coaching support; dCBTi with virtual coaching; dCBTi without coaching
Behavioral: Virtual coaching — A virtual coach will be added to the app functionality. It will be in the form of a text-based forced-choice conversation bot. It will initiate conversations with the users to check their understanding of treatment materials and guide them to come up with specific action plans to implement the treatment strategies.
  Arms: dCBTi with non-therapist coaching support; dCBTi with therapist coaching support; dCBTi with virtual coaching
Behavioral: Non-therapist coaching — A research intern will answer questions and address concerns raised by the participant at the end of modules 1, 3, and 6 by phone. The contact time will be within 30 minutes on each occasion.
  Arms: dCBTi with non-therapist coaching support
Behavioral: Therapist coaching — A clinical psychology trainee will provide therapeutic support to enhance the use and adherence to CBTi treatment strategies at the end of modules 1, 3, and 6 by phone. The contact time will be within 30 minutes on each occasion.
  Arms: dCBTi with therapist coaching support
Behavioral: Sleep Hygiene and Self-Monitoring Control — An app with self-monitoring function and videos and written materials about sleep hygiene will be provided.
  Arms: Digital Sleep Hygiene and Self-Monitoring Control

SUMMARY:
The current research aims to evaluate the adherence and efficacy of dCBTi with different types of coaching support.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of the five conditions. C1: Sleep Hygiene and Self-Monitoring Control Condition; C2: dCBTi without coaching; C3; dCBTi with virtual coaching; C4: dCBTi with non-therapist coaching; C5: dCBTi with therapist coaching.

Question 1:

Does dCBTi work better than the active control?

Hypothesis 1:

Participants in C2, C3, C4, and C5 will have greater improvement in insomnia than those in C1.

Question 2:

Does coaching support, virtual or human, improve treatment adherence and outcome?

Hypothesis 2:

Participants in C3, C4, and C5 will have greater improvement in insomnia and greater adherence to treatment recommendations than those in C2.

Question 3:

Does human coaching enhance treatment adherence and outcome?

Hypothesis 3:

Participants in C4 and C5 will have greater improvement in primary outcome than those in C3.

Question 4:

Does therapist-coaching-support enhance treatment adherence and outcome to a greater extent than virtual and non-therapist coaching support?

Hypothesis 4:

Participants in C5 will have greater improvement in primary outcome than those in C3 and C4.

ELIGIBILITY:
Inclusion Criteria:

* (a) Hong Kong resident,
* (b) Aged 18 or above,
* (c) Able to read and write Chinese,
* (d) Has regular access to a smart phone and internet,
* (e) insomnia severity index ⩾10;
* (f) Willing and can be contacted by experimenter via phone between 9 am - 9 pm

Exclusion Criteria:

* (a) significant untreated/unstable mental or medical illness,
* (b) known factor to interfere with participation in this research,
* (c) serious medical, neurological, or psychiatric illness that may affect participation in this research,
* (d) sleep apnea,
* (e) concurrent treatment for insomnia,
* (f) unstablized medication that can affect sleep

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Insomnia Severity Index (ISI) | 12 weeks from baseline
  Insomnia symptoms measured by the Insomnia Severity Index (ISI). The score ranges from 0 to 24. Higher scores indicate greater levels of insomnia symptoms

SECONDARY OUTCOMES:
Changes in Sleep Condition Indicator (SCI) | 12 weeks from baseline
  Insomnia symptoms measured by the Sleep Condition Indicator (SCI). The score ranges from 0 to 32. Higher scores indicate lower levels of insomnia symptoms
Changes in sleep efficiency | 12 weeks from baseline
  Sleep efficiency measured by Consensus Sleep Diary. It ranges from 0 to 100%, the higher indicates better sleep
Changes in sleep onset latency (SOL) | 12 weeks from baseline
  Sleep onset latency (SOL) measured by Consensus Sleep Diary. Its unit is minutes. Longer SOL indicates greater levels of insomnia
Changes in wake after sleep onset | 12 weeks from baseline
  Wake after sleep onset (WASO) measured by Consensus Sleep Diary. Its unit is minutes. Longer WASO indicates greater levels of insomnia
Changes in sleep-related cognitions | 12 weeks from baseline
  Sleep-related cognitions measured by the Dysfunctional Beliefs and Attitudes about Sleep 16-item Scale (DBAS-16). Respondents rate their agreement to each of the 16 statements on a Visual Analog Scale (0-100). Higher scores indicate more dysfunctional sleep-related cognitions.
Changes in sleep-related safety behaviors | 12 weeks from baseline
  Sleep-related safety behaviors measured by the Sleep-Related Behavior Questionnaire - 20 (SRBQ-20). The score ranges from 0 to 80, higher scores indicate greater engagement in sleep-related safety behaviors
Changes in daytime sleepiness | 12 weeks from baseline
  Sleepiness measured by the Epworth Sleepiness Scale (ESS). The score ranges from 0 to 24, higher scores indicate greater sleepiness.
Changes in fatigue | 12 weeks from baseline
  Fatigue measured by the Fatigue Assessment Scale (FAS). The score ranges from 10 to 50, the higher the greater levels of fatigue
Changes in depressive symptoms | 12 weeks from baseline
  Depressive symptoms measured by the Patient Health Questionnaire - 9 (PHQ-9). The score ranges from 0 to 27, the higher the more depressed
Changes in anxiety symptoms | 12 weeks from baseline
  Anxiety symptoms measured by the Generalized Anxiety Disorder 7-item Scale (GAD-7). The score ranges from 0 to 21, the higher the more anxious
Changes in psychological wellbeing | 12 weeks from baseline
  Psychological wellbeing measured by the Satisfaction with Life Scale (SWLS). The score ranges from 5 to 35, the higher indicates greater wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sze Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available for sharing with other researchers for secondary analysis upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From after the study findings have been published to 5 years afterwards.
Access Criteria: The request party has a pre-registration of the research that requires data from the present study indicating clearly what data are required and other criteria as the PI deem appropriate.

REFERENCES:
- [Derived] Chan WS, Cheng WY, Lok SHC, Cheah AKM, Lee AKW, Ng ASY, Kowatsch T. Assessing the Short-Term Efficacy of Digital Cognitive Behavioral Therapy for Insomnia With Different Types of Coaching: Randomized Controlled Comparative Trial. JMIR Ment Health. 2024 Aug 7;11:e51716. doi: 10.2196/51716. PMID 39110971